CLINICAL TRIAL: NCT01087684
Title: A Prospective, Randomized, Clinically Based Study on the Response to Selective Laser Trabeculoplasty Versus Argon Laser Trabeculoplasty in Patients Who Are Under 60 Years of Age
Brief Title: Response to SLT vs. ALT in Patients Under 60 Years of Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Catherine Birt, MD, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 459-2004
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Glaucoma
Keywords: Glaucoma; laser trabeculoplasty; intraocular pressure
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Argon laser trabeculoplasty (Active Comparator): Patients received standard argon laser treatment
  Interventions: Procedure: Argon laser trabeculoplasty
- Selective laser trabeculoplasty (Active Comparator): Patients received a standard selective laser treatment
  Interventions: Procedure: Selective laser trabeculoplasty

INTERVENTIONS:
Procedure: Argon laser trabeculoplasty — Argon laser 600-800 mW, 0.1seconds, 50 micron spot size, 45 - 55 burns over 180 degrees of trabecular meshwork
  Other Names: ALT
  Arms: Argon laser trabeculoplasty
Procedure: Selective laser trabeculoplasty — Selective laser trabeculoplasty 0.7 - 0.8 mJ, 400 micron spot size, 3 nanosecond, 45 - 55 burns over 180 degrees of trabecular meshwork.
  Other Names: SLT
  Arms: Selective laser trabeculoplasty

SUMMARY:
Laser trabeculoplasty is a routine treatment for glaucoma and can be performed with either argon (ALT) or selective Yag (SLT) lasers. The effectiveness of each has not been studied in patients under 60 years, which is younger than average for the procedure. The study hypothesis is that there will be no difference between the two laser types.

DETAILED DESCRIPTION:
Forty-two young patients (age 29 to 60) had one eye randomized to ALT (n = 22) or SLT (n = 20). Intraocular pressure was measured prior to laser and 1 hour, 1 day, 6 weeks, 3 months, every 3 months until 2 years, and then yearly post-laser. χ2 analysis and student's t-test were used to determine statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Age < 60 years
* Intraocular pressure not adequately controlled

Exclusion Criteria:

* Prior laser treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2004-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | Two years
  The intraocular pressure was measured at 6 weeks, 4.5 months, 9, 12, 18 and 24 months following the laser treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine M Birt, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Result] Liu Y, Birt CM. Argon versus selective laser trabeculoplasty in younger patients: 2-year results. J Glaucoma. 2012 Feb;21(2):112-5. doi: 10.1097/IJG.0b013e318202791c. PMID 21572334